CLINICAL TRIAL: NCT02694107
Title: A Randomized Controlled Trial of Effectiveness of Proprioceptive Training on Dynamic Postural Balance During Pregnancy
Brief Title: Effectiveness of Proprioceptive Training on Dynamic Postural Balance During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Fayiz Elshamy, Faculty of physical therapy, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FF1972
Record Dates: First submitted 2016-02-01; First posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Disturbance; Balance; Pregnancy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proprioceptive exercises (Experimental): Proprioceptive exercises performed 3 sessions per week for 4weeks
  Interventions: Other: Proprioceptive exercises; Other: Control
- Control (No Intervention): Without any exercises

INTERVENTIONS:
Other: Proprioceptive exercises
  Arms: Proprioceptive exercises
Other: Control
  Arms: Proprioceptive exercises

SUMMARY:
The purpose of the present study was to measure the effect of proprioceptive training, short-term, on dynamic postural balance during pregnancy and after 8 weeks of follow-up.

Thirty-nine pregnant women were randomized to either the intervention group(n=20) , which would perform proprioceptive exercise, or the control group(n=19, no intervention) .

DETAILED DESCRIPTION:
Improvement in the postural balance of pregnant women may be the improvement in joint mechanoreceptor activation present in the joint capsules, medial ligament, posterior cruciate ligament, and meniscus, which result in improved articular stabilization and, consequently, a possible increase in the musculature's ability to provide co-contraction.

Improved their postural control after the intervention may have been due to central and peripheral nervous system balance control circuits and strength gains, which showed improvements extending from the second to the third trimester . The maintenance of postural balance requires the integration of the visual, vestibular, and somatosensory systems.

At the spinal level, first level of motor control, nervous reflex movement patterns are received from higher levels of the nervous system. This provides for reflex splinting during conditions of abnormal stress about the joint and has significant implications for rehabilitation.The muscle spindles play a major role in the control of muscular movement by adjusting activity in the lower motor neurons.

The second level of motor control is the brain stem, where the joint afferent is relayed to maintain the posture and balance of the body. Information delivered to the brain stem emanates from the joint proprioceptors, the vestibular centers in the ears, and the eyes.The final aspect of motor control includes the highest level of CNS function (motor cortex, basal ganglia, and cerebellum)and is mediated by cognitive awareness of body position and movement. Movements that are repeated can be stored as central commands, and can be performed without continuous reference to consciousness. This better joint afferent between the peripheral and central nervous system control may be reflected in the improvement of balance during pregnancy, as observed in this study as a result of proprioceptive training delivered to pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age between 25 and 30 years,
* Gestational age was 20 weeks gestation,
* Body mass index not exceeding 30 kg/m2,
* Low risk pregnancy,
* Single fetus,
* Healthy sensory motor function in the lower limbs.

Exclusion Criteria:

* Gestational diabetes,
* Pre-eclampsia,
* Toxemia,
* Gestational hypertension,
* Previous abortion,
* High-risk pregnancy,
* Type I or Type II diabetes ,
* Any condition that could affect sensation,
* A leg or foot fracture or ankle or knee sprain within the last year,
* Current back or knee pain,
* Cardiovascular, neurologic, neuromuscular, or pulmonary disease,
* Vertigo, balance or any visual problems,or psychological illness.
* Current smokers,
* Currently taking any medication that would affect their ability to balance.

Ages: 25 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Anteroposterior (AP), mediolateral (ML), and global postural sway(GPS) indices were measured at 20 weeks gestation | up to 20 weeks
  Dynamic balance(AP,ML and GPS) indices were measured by the Biodex Balance System at 20 weeks gestation(WG).
Anteroposterior (AP), mediolateral (ML), and global postural sway(GPS) indices were measured at 24 weeks gestation | up to 24 weeks
  Dynamic balance(AP,ML and GPS) indices were measured by the Biodex Balance System at 24 weeks gestation(WG).
Anteroposterior (AP), mediolateral (ML), and global postural sway(GPS) indices were measured at 32 weeks gestation | up to 32 weeks
  Dynamic balance(AP,ML and GPS) indices were measured by the Biodex Balance System at 32 weeks gestation(WG).

CONTACTS AND LOCATIONS:
Overall Officials: Ana Paula Ribeiro, Prof. Dr, Study Chair — Department of Physical Therapy, Laboratory of Biomechanics and Rehabilitation Musculoskeletal, University of Santo Amaro and Researcher at the University of São Paulo, São Paulo, Brazil.

IPD SHARING:
Plan to Share IPD: No